CLINICAL TRIAL: NCT06919146
Title: A 12-week Afterschool Game-Based Physical Activity Program Improves Physical Fitness of 9-10-Year-Old Children: A Randomized Controlled Study
Brief Title: After-school Game-Based Physical Activity Program Improves Physical Fitness of 9-10-Year-Old Children
Acronym: AGPAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Elvin Onarici Gungor (Other)
Responsible Party: Sponsor-Investigator, Elvin Onarici Gungor, Principal Investigator, Eskisehir Technical University
Organization: Eskisehir Technical University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: EskisehirTU-SBF-EOG-01; Eskisehir Technical University (Other: Education)
Record Dates: First submitted 2025-03-12; First posted 2025-04-09 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Physical Activity
Keywords: Game; Physical activity; Afterschool program; Physical fitness
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: The study was a parallel-group, a simple randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental Group (Experimental): EG additionally participated in AGPAP (4:00 pm-5:00 pm) twice a week, every Wednesday and Friday, for a total of 60 minutes, for 12 weeks. AGPAP started the week after the pre-tests for EG. The intervention program consisted of 24 traditional street games, including running, hopping, galloping, leaping, jumping, sliding, striking, catching, ball catching, overhand throwing, balance, one-hand throwing, flexibility, coordination, shooting at the target, and hand-arm-leg strength and both outdoor and indoor facilities were utilized based on whether conditions. Each practice phase is 60 minutes long and includes three stages: instruction and warm-up (10 min.), AGPAP practice (45 min.), and cooling-down (5 min.). Two researchers who hold graduate degrees in physical education and sport led AGPAP and recorded children's participation. At the end of the intervention, the same testing procedures and testing materials were used for post-test measurements.
  Interventions: Behavioral: Physical Activity
- Control (No Intervention): Measurements were applied to the CG

INTERVENTIONS:
Behavioral: Physical Activity — EG participated in AGPAP (4:00 pm-5:00 pm) twice a week, every Wednesday and Friday, for a total of 60 minutes, for 12 weeks. EG and CG did not participate in any additional physical activity programs after-school.
  Arms: Experimental Group

SUMMARY:
This study investigates the effect of an afterschool game-based physical activity program (AGPAP) on children's PF. This study was randomized controlled trial involving 120 children from a state school in Eskisehir/Turkey. The CONSORT checklist was used in this study. The sample of 9-10 years children (n = 120) was divided into groups by randomization. The intervention consisted of AGPAP. For PF, handgrip strength, curl-ups, sit-and-reach, standing long jump, and 10-meter running speed tests were applied.

ELIGIBILITY:
Inclusion Criteria:

1. being 9-10-year-old,
2. volunteering,
3. permission from the child's parents,
4. not having any amputations or permanent disabilities in their bodies,
5. not having chronic or acute diseases,
6. not using a support device.

Exclusion Criteria:

1. any discomfort during measurements,
2. the child does not want to participate in the measurement,
3. the child does not participate in the practices due to any disability or discomfort,
4. not reaching 80% participation in the program.

Ages: 9 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 130 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2020-08-27 (Actual); Study Completion 2020-12-07 (Actual)

PRIMARY OUTCOMES:
Body Mass Index | 12 weeks
  Body weights were measured using a digital scale (SECA, Hamburg) with an accuracy of 0.1 kg while subjects were wearing as light clothing as possible and barefoot. Heights were measured using a portable stadiometer (SECA, Hamburg) with an accuracy of 0.1 cm while subjects were barefoot, with their feet together and their heads on a horizontal plane 47. The weight(kg)/height2(m) formula was used to calculate BMI.

SECONDARY OUTCOMES:
Handgrip strength test | 12 weeks
  The hand grip strength test measures the explosive power of the upper body using an adjustable and calibrated hand dynamometer (Takei, Tokyo, Japan). Participants were asked to hold them in their right and left hands and squeeze it slowly and continuously until they reached the max. for at least 2 s. The best of 2 repetitions was recorded as the test score in kg.
Standing long jump test | 12 weeks
  Each participant attempted to jump as far as possible across a certain distance while standing, with their arms forward, their feet closed, and landing on the ground. The best of the 2 attempts was recorded in centimeters.
Curl-ups test | 12 weeks
  Participants were asked to lie with their arms crossed on their chest, their knees bent, and their feet flat on the floor. Afterward, they were asked to lift their upper bodies with their elbows facing forward, touch their knees, and then return to the lying position. The total number of complete curl-ups performed correctly in 30 seconds was recorded.
The sit and reach test | 12 weeks
  The sit and reach tests were applied using a specially constructed box that had a slide runner attached to the top. The accuracy of the instrument used was 0.1 cm, and the length it was able to measure was 80 cm (01285A, Lafayette, USA). Subjects sat on a flat surface with their back, shoulders, and the back of their head close to the wall for the sit-and-reach test. Their arms were straightened, their hands were placed on the tester board with palms facing down, and their legs were positioned straight. Each participant placed their hands side by side on the measurement starting line on the bench and gradually pushed the bar on the sit-and-reach bench forward to the furthest point they could while reaching with their hands without bending their knees. Each participant repeated the test two times, and the best of these two repetitions was taken into statistical evaluation.
10-meter running speed test | 12 weeks
  Photocells were placed at the beginning and end of the 10-meter track (Smart Speed, Fusion Sport, Brisbane, Australia). Participants waited in a standing starting position 50 cm behind the starting line and started sprinting upon receiving the command when they were ready. Two repetitions were conducted, and the best result was recorded at the end of the trials.

CONTACTS AND LOCATIONS:
Overall Officials: ELVİN ONARICI GÜNGÖR, dr, Principal Investigator — ESKISEHIR TECNICAL UNIVERSITY
Locations (1):
- Eskisehir Tecnical University, Odunpazari, Eskişehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
only IPD used in the results publication
Supporting Information: Study Protocol, ICF
Time Frame: January 2025-January 2026

REFERENCES:
- [Derived] Onarici Gungor E, Yaliz Solmaz D, Guven G, Gurol B. A 12-week afterschool game-based physical activity program improves physical fitness of 9-10-year-old children: a randomized controlled study. Sci Rep. 2025 Dec 4;15(1):44013. doi: 10.1038/s41598-025-31429-9. PMID 41345233